CLINICAL TRIAL: NCT06403254
Title: Seeking Bacterial Prevalence for Targeted Pre-Surgical Antibiotic Prophylaxis in Prosthetic Surgery
Brief Title: Evaluation of VSS Antibiotic Prophylaxis in Prosthetic Surgery (MRSA)
Acronym: MRSA
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: MRSA
Record Dates: First submitted 2024-01-26; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-02

CONDITIONS: Infection in Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: There isn't an intervention name because the study is observational and has only one group. — Follow-up after surgey

SUMMARY:
based on international guide lines, antibiotic prophylaxis in Orthoaedic major surgery has to be done with a Cephalosporin 1st generation (e.g. Cefazolin 1 g 30' before surgery).

Since more than 10 years ago the investigators started evaluatinf infections in such a surgery, well demosntrating a level below 1% and, more important, a responsability of MRSA. considering Cephalosporin 1st generation useful but not determinat in such a surgery, investigators consider the use of a Glycopepide (Vancocyn 1 g in Very short. The primary outcome is to evaluate the validity of such proposal, performing a study of prevalence.

DETAILED DESCRIPTION:
Patients enrolled in the study have to follow rhese steps:

T0: Clinical evaluation and Cephalosporin VSS prophylaxis, as usual T1: Surgery for TKA or THA T2: Post-operative --> control and, if an infextion is supposed, Coltural examination and ABG T3: Post-op orthopedic control at 6 months, to evaluate any possible infection T4: Post-op clinical valuation at 12 months, with the same goal

ELIGIBILITY:
Inclusion Criteria:

Patiens male and female, old more than 40 years TKA or THA Surgeryntervento di chirurgia protesica ASAC II or even III, without any acute coexisting disease Informed consent -

Exclusion Criteria:Patients with infection before surgery Immunocompromise patient (e.g. Diabeties with glicate HB indicating a metabolic bad compensation) Patient with coagulation disorders Pregnancy Informed consent denied

-

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients, in a consecutive serie, based on criteria over indicated
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Infections | 1 year after the surgery
  Orthopedic clinical control , with or without exams

CONTACTS AND LOCATIONS:
Locations (1):
- Istitutio Ortopedico Galeazzi Sede San Siro, Milan, Lumbardy, Italy

IPD SHARING:
Plan to Share IPD: No